CLINICAL TRIAL: NCT01459952
Title: A Double-blind, Randomised, Parallel Group, Phase III Comparative Study With Rose-hip Liquid and Placebo Given to Healthy Volunteers in the Winter Season Aiming to Evaluate the Occurences of Flu and Catching a Cold
Brief Title: A Double-blind, Randomised, Parallel Group,Comparative Study With Rose-hip Liquid and Placebo Given to Healthy Volunteers in the Winter Season Aiming to Evaluate the Occurences of Flu and Catching a Cold
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hyben Vital ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HV 02/11
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Flu; Common Cold
Keywords: occurences of flu; occurences of common cold
MeSH Terms: conditions — Influenza, Human; Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rose hip Liquid (Experimental): 20 ml Rose hip Liquid BID
  Interventions: Dietary Supplement: Rose hip Liquid
- Placebo (Placebo Comparator): 20 ml placebo liquid BID
  Interventions: Dietary Supplement: Rose hip Liquid

INTERVENTIONS:
Dietary Supplement: Rose hip Liquid — Rose hip Liquid, 20 ml BID

SUMMARY:
The trial is an investigator-initiated, double-blind, randomized, placebo-controlled phase III study.

After the patient has receiving information about the study and after given written informed consent, the patient will be screened.

The patient's medical history and demographic information will be recorded. The patient will then be asked questions in accordance to the study questionnaires, and they will also be asked to complete questionnaires regarding quality of life - and finally they be instructed on how to complete the diary.

All patients are randomized to receive standardized rose hip liquid or matching placebo. The subject is instructed to take the liquid form of rose hips in the morning and evening meal. The subject will also be advised to call the clinic if there is an acute attack of cold and / or flu because they must then increase the in-take of study treatment to 3 double dose for 5 days and then return to normal dose.

The subject will then be asked a series of questions under study questionnaires, and be instructed in how questionnaires (SF-12) and diary filled. This is to provide security to the validation output values Investigator or study nurse will take telephone contact with the subject once a month, subjects will be asked about how things are going and to remember to take the liquid and whether they have completed the diary.

The last patient visit will take place after 6 months. Any side effects will be reported to and reviewed with HybenVital ApS in collaboration with medical experts.

ELIGIBILITY:
Inclusion Criteria:

* First Men and women aged 50 + years
* It is accepted that the subjects can be treated for medical diseases.
* It is also accepted that the subjects receiving daily medication such as diuretics and medication for Hypertension, hypercholesterolemia and blood glucose-lowering treatment, medicine that strengthens the heart, symptom-relieving medication for joint disease, etc.
* Subjects may also use n-3 fatty acids (fish oil), as long as the fixed dosage.

Exclusion Criteria:

* Subjects who have been treated with rose hip extracts or powder within 3 months before screening.
* Subjects who have been treated with ginger, avocado / soy, large doses of vitamins (including vitamin C) or other known dietary supplements within 3 months before screening
* Subjects that have been deemed to be have a hard time collaboration
* Subjects who abuse narcotics.
* Subjects who abuse alcohol
* Subjects with a current mental illness
* Subjects with known allergy to rose hips
* Subjects participating in another clinical trial, or have participated in another clinical trial within 3 months before this trial started.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Frequency and duration of colds and flu attacks | 6 months
  Frequency and duration of colds and flu attacks will be analyzed within each of the two treatments (Rose hip Liquid and Placebo). The severity will also be assessed by recording the intensity of coughing, how much pain the patient has felt in the throat and if there is fever, headache and / or fatigue

SECONDARY OUTCOMES:
Quality of life | 6 months
  Quality of life by SF-12 will be assessed within each group in what is seen on the initial value vs. the final value at study end, and the difference between active and placebo.
Sleep quality | 6 months
  General wellbeing concerning sleep quality. Measured by using entries in the patient diary: Baseline vs.6 months and active treatment vs. placebo treatment
Pain in muscles and joints | 6 months
  General wellbeing concerning pain in muscles and joints. Measured by using entries in the patient diary: Baseline vs.6 months and active treatment vs. placebo treatment
Stiffness in muscles and joints | 6 months
  General wellbeing concerning stiffness in muscles and joints. Measured by using entries in the patient diary: Baseline vs.6 months and active treatment vs. placebo treatment
Body weight | 6 months
  Weight changes seen at Baseline vs.6 months and active treatment vs. placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kaj Winther, Dr, Principal Investigator — Department of clinical biochemical
Locations (1):
- Frederiksberg University Hospital, Frederiksberg, Denmark